CLINICAL TRIAL: NCT00158301
Title: Continuation Phase CBT for Youth With MDD
Brief Title: Cognitive Behavioral Therapy for Depression Relapse Prevention in Children and Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Beth Kennard, PsyD, UT Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R34MH072737 (NIH); R34MH072737 (NIH); DSIR 84-CTS
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-11

CONDITIONS: Depression
Keywords: Child; Adolescent; CBT; Drug Therapy
MeSH Terms: conditions — Depression | interventions — Cognitive Behavioral Therapy; Drug Therapy; Fluoxetine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Continuation phase cognitive behavioral therapy and drug therapy for 6 more months following acute treatment response
  Interventions: Behavioral: Cognitive behavioral therapy (CBT); Drug: Drug therapy
- 2 (Active Comparator): Continuation phase drug therapy only for 6 more months following acute treatment response
  Interventions: Drug: Drug therapy

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy (CBT) — CBT sessions will focus on teaching participants skills to manage depressed moods and to identify situations which might put them at risk for a relapse in depressive symptoms.
  Arms: 1
Drug: Drug therapy — All participants will receive 12 weeks of treatment with antidepressant therapy. Responders to initial treatment will continue medication during the continuation phase (both treatment arms).
  Other Names: fluoxetine

SUMMARY:
This study will determine the effectiveness of cognitive behavioral therapy in preventing a relapse of depressive symptoms in children.

DETAILED DESCRIPTION:
Depression is a chronic and episodic condition that may have devastating effects on social and emotional functioning, particularly in the pediatric population. While approximately 90% of children eventually recover from an episode of depression, up to 40% of those children relapse within 1 to 2 years. Data indicate that cognitive behavioral therapy (CBT) delivered after depressive symptoms subside can significantly reduce depression relapses in adults. However, there are no comparable studies in children or adolescents. This study will determine whether CBT is effective in reducing a relapse of depressive episodes in children and adolescents with major depression.

This study comprises two phases. In Phase 1, all participants will receive drug treatment for 12 weeks. Participants who respond to the treatment will complete the study after 12 weeks. Participants whose depression symptoms return after 12 weeks will be enrolled in Phase 2. In Phase 2, participants will be randomly assigned to either continue drug therapy alone or to receive drug therapy plus CBT for 6 months. The CBT will focus on teaching participants skills to manage depressed moods and to identify situations which might put them at risk for a relapse in depressive symptoms. Self-report scales will be used to assess the depressive symptoms of participants who complete Phases 1 and 2 at study entry and at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of nonpsychotic major depressive disorder at least 4 weeks prior to study entry
* Clinical Global Impression severity score of 4 or greater
* Children's Depression Rating Scale score of 40 or greater
* Currently attending school
* Willing and able to use acceptable methods of contraception, if applicable
* In good general health
* Parent or guardian willing to provide informed consent, if applicable

Exclusion Criteria:

* History of psychotic disorders
* Alcohol or substance abuse or dependence within 6 months prior to study entry
* History of anorexia nervosa or bulimia
* Chronic medical illness requiring regular medication
* Current use of medication with psychotropic effects
* First-degree relatives (e.g., mother, father, sister, brother) with bipolar I disorder
* At risk for suicide
* Failure of a previous adequate treatment with fluoxetine (defined as at least 40 mg/day for 4 weeks)
* IQ less than 80
* Pregnancy or breastfeeding

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72 (Actual)
Dates: Start 2004-09; Primary Completion 2007-11 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Relapse of depressive symptoms | Measured at Months 3 and 9

CONTACTS AND LOCATIONS:
Overall Officials: Beth D. Kennard, PsyD, Principal Investigator — University of Texas, Southwestern Medical Center at Dallas
Locations (1):
- University of Texas Southwestern Medical Center at Dallas, Dallas, Texas, United States

REFERENCES:
- [Derived] Nakonezny PA, Hughes CW, Mayes TL, Sternweis-Yang KH, Kennard BD, Byerly MJ, Emslie GJ. A comparison of various methods of measuring antidepressant medication adherence among children and adolescents with major depressive disorder in a 12-week open trial of fluoxetine. J Child Adolesc Psychopharmacol. 2010 Oct;20(5):431-9. doi: 10.1089/cap.2009.0108. PMID 20973714
- [Derived] Kennard BD, Emslie GJ, Mayes TL, Nightingale-Teresi J, Nakonezny PA, Hughes JL, Jones JM, Tao R, Stewart SM, Jarrett RB. Cognitive-behavioral therapy to prevent relapse in pediatric responders to pharmacotherapy for major depressive disorder. J Am Acad Child Adolesc Psychiatry. 2008 Dec;47(12):1395-404. doi: 10.1097/CHI.0b013e31818914a1. PMID 18978634